CLINICAL TRIAL: NCT06667245
Title: Impact on Quality of Life and Burden of Disease in Adults With Herpes Zoster
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: V1.0_03.04.24
Record Dates: First submitted 2024-07-09; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Herpes Zoster; Quality of Life; Immunization; Infection
MeSH Terms: conditions — Herpes Zoster; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients > 18 years old who are going to be immunized against HZ: Patients > 18 years old who are going to be immunized against HZ

SUMMARY:
Title: Impact on quality of life and disease burden in adults with herpes zoster

Prospective cohort study for the primary objective and the secondary objectives (1 and 2) and retrospective cohort study for the secondary objective 3.

Disease or disorder under study: Patients with a herpes zoster (HZ) diagnosis.

DETAILED DESCRIPTION:
Impact on quality of life and disease burden in adults with herpes zoster Contents

HYPOTHESIS AND OBJECTIVES OF THE STUDY 3.1 Hypothesis: Herpes zoster significantly affects the quality of life of those who suffer from it with a high disease burden.

3.2 Primary outcomes: To measure the quality of life of patients with a history of herpes zoster who attend the immunization unit of the Fundación Jiménez Díaz University Hospital.

3.3 Secondary outcomes

1. Evaluating the quality of life according to the location of the zoster (postherpetic neuralgia, ophthalmic zoster, etc.)
2. Evaluating the effectiveness of the vaccine against herpes zoster in terms of number of episodes, severity and quality of life.
3. Evaluating the economic impact and disease burden in terms of morbidity and mortality in adult with herpes zoster

TYPE OF STUDY AND DESIGN

Prospective cohort study for the primary objective and the secondary objectives (1 and 2) and retrospective cohort study for the secondary objective 3.

Disease or disorder under study: Patients with a herpes zoster (HZ) diagnosis.

SUBJECT SELECTION 5.1 Prospective cohort study Inclusion criteria Patients > 18 years of age who are to be immunised against HZ

Exclusion criteria:

* Pregnant women
* Patients with altered level of consciousness (dementia and others) who do not complete the questionnaires
* Patients who do not wish to participate in the study 5.2 Retrospective cohort study Inclusion criteria
* Adults over 18 years of age with a diagnosis of HZ in the CMBD from 2012 to 2023 at the Jiménez Díaz Foundation. Since the international classification of diseases changed from ICD 9 to ICD 10 in 2016, the codes to be used for the inclusion of patients in the study are described below.

ICD 9 053 Herpes zoster Includes:

Herpes zoster Zone 053.0 With meningitis 053.1 With other central nervous system complications 053.10 With unspecified nervous system complications 053.11 Geniculate herpes zoster or Herpetic geniculate ganglionitis 053.12 Postherpetic trigeminal neuralgia 053.13 Postherpetic polyneuropathy 053.14 Herpes zoster myelitis 053.19 Other 053.2 With ophthalmic complications 053.20 Herpes zoster dermatitis of eyelid or Herpes zoster ophthalmicus 053.21 Herpes zoster keraconjunctivitis 053.22 Herpes zoster iridocyclitis 053.29 Other 053.7 With other complications specific 053.71 Otitis externa due to herpes zoster 053.79 Other 053.8 With unspecified complications 053.9 Herpes zoster without complication Herpes zoster NOS ICD 10 B02 Herpes zoster Includes: - herpes - zone B02.0 Encephalitis due to herpes zoster Meningoencephalitis due to herpes zoster B02.1 Meningitis due to herpes zoster B02.2 Herpes zoster with other nervous system involvement B02.21 Postherpetic geniculate ganglionitis B02.22 Postherpetic trigeminal neuralgia B02.23 Postherpetic polyneuropathy B.02.24 Postherpetic myelitis or Herpes zoster myelitis B02.29 Other postherpetic nervous system involvement or Postherpetic radiculopathy B02.3 Ocular herpes zoster B02.30 Ocular herpes zoster, unspecified B02.31 Herpes zoster conjunctivitis B02.32 Herpes zoster iridocyclitis B02.33 Herpes zoster keratitis or Herpes zoster keratoconjunctivitis B02.34 Herpes zoster scleritis B02.39 Other herpes zoster eye diseases or Herpes zoster blepharitis B02.7 Disseminated herpes zoster B02.8 Herpes zoster with other complications Herpes zoster otitis externa B02.9 Uncomplicated herpes zoster Herpes zoster

ELIGIBILITY:
1 Prospective cohort study Inclusion criteria Patients > 18 years of age who are to be immunized against HZ

Exclusion criteria:

* Pregnant women
* Patients with altered level of consciousness (dementia and others) who do not complete the questionnaires
* Patients who do not wish to participate in the study 5.2 Retrospective cohort study Inclusion criteria Adults >18 years of age with a diagnosis of HZ in the CMBD from 2012 to 2023 at the Jiménez Díaz Foundation hospital. Since the international classification of diseases changed from ICD 9 to ICD 10 in 2106, the codes to be used for the inclusion of patients in the study are described below.

ICD 9 053 Herpes zoster

Includes:

* Herpes zoster
* Zone 053.0 With meningitis 053.1 With other central nervous system complications
* 053.10 With unspecified nervous system complications
* 053.11 Geniculate herpes zoster or Herpetic geniculate ganglionitis
* 053.12 Postherpetic trigeminal neuralgia
* 053.13 Postherpetic polyneuropathy
* 053.14 Herpes zoster myelitis
* 053.19 Other 053.2 With ophthalmic complications
* 053.20 Herpes zoster dermatitis of eyelid or Herpes zoster ophthalmicus
* 053.21 Herpes zoster keratoconjunctivitis
* 053.22 Herpes zoster iridocyclitis zoster
* 053.29 Other 053.7 With other specific complications
* 053.71 Otitis externa due to herpes zoster
* 053.79 Other 053.8 With unspecified complications 053.9 Herpes zoster without complication Herpes zoster NOS ICD 10 B02 Herpes zoster

Includes:

* herpes
* zona B02.0 Encephalitis due to herpes zoster Meningoencephalitis due to zoster B02.1 Meningitis due to herpes zoster B02.2 Herpes zoster with other nervous system involvement
* B02.21 Postherpetic geniculate ganglionitis
* B02.22 Postherpetic trigeminal neuralgia
* B02.23 Postherpetic polyneuropathy
* B.02.24 Myelitis Postherpetic myelitis
* B02.29 Other postherpetic nervous system involvement
* B02.3 Ocular herpes zoster
* B02.30 Ocular herpes zoster, unspecified
* B02.31 Herpes zoster conjunctivitis
* B02.32 Herpes zoster iridocyclitis
* B02.33 Herpes zoster keratitis
* B02.34 Herpes zoster scleritis
* B02.39 Other herpes zoster eye disease
* B02.7 Disseminated herpes zoster
* B02.8 Herpes zoster with other complications
* B02.9 Uncomplicated herpes zoster
* B02.39 Herpes zoster otitis externa NEOM

Exclusion criteria:

Patients who are vaccinated against HZV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective study:
  Patients > 18 years of age who are to be immunized against HZ
  Retrospective study:
  Adults over 18 years of age with a diagnosis of HZ in the CMBD from 2012 to 2023 at the Jiménez Díaz Foundation hospital.
  Since the international classification of diseases changed from ICD 9 to ICD 10 in 2016, the codes to be used for the inclusion of patients in the study are described below.
  Patients diagnosed with herpes zoster (HZ). Study Population and Total Number of Patients: Based on the sample calculation, it is intended to include a total of 357 patients in the prospective study and 1,920 patients in the retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 357 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-11-04 (Estimated); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patients with a history of herpes zoster who attend the immunization unit of the Jiménez Díaz Foundation University Hospital. | Data will be collected for 1 year and then analyzed to respond to the outcomes
  Measuring the quality of life of patients with a history of herpes zoster who attend the immunization unit of the Jiménez Díaz Foundation University Hospital.

SECONDARY OUTCOMES:
Quality of life according to the location of herpes zoster | Data will be collected for 1 year and then analyzed to respond to the outcome
  Evaluate quality of life according to the location of herpes zoster (postherpetic neuralgia, ophthalmic zoster, etc.)
Effectiveness of the vaccine against herpes zoster | Data will be collected for 1 year and then analyzed to respond to the objective
  Evaluating the effectiveness of the herpes zoster vaccine in terms of the number of episodes, severity and quality of life.
Economic impact and disease burden in terms of morbidity and mortality | A retrospective analysis will be carried out, when the data has been analysed this outcome will be answered, in approximately 6 months.
  Economic impact and burden of disease in terms of morbidity and mortality of adult patients with herpes zoster

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Patil A. Goldust M. Wollina U. Herpes zoster: A Review of Clinical Manifestations and Management. Viruses. [Internet]. 2022. [Consultado 18 Feb 2024]; 14(2) — https://pubmed.ncbi.nlm.nih.gov/35215786/
- See also: Kain A., Tizek L., Wecker H., Wallnöfer F., Biedermann T., Zink A. Evaluating public interest in herpes zoster in Germany by leveraging the internet: a retrospective search data analysis. BMC Public Health. [Internet]. 2023. [Consultado 29 Mar 2024]; 2 — https://pubmed.ncbi.nlm.nih.gov/37580664/
- See also: Masa Calles J. López Perca N. Vila Cordero B. Carmona R. Vigilancia y epidemiología del herpes zóster en España. RevEsp Salud Pública.[Internet]. 2021. [Consultado 18 Feb 2024]; 95. (e1-13). — https://www.sanidad.gob.es/biblioPublic/publicaciones/recursos_propios/resp/revista_cdrom/VOL95/ORIGINALES/RS95C_202106088.pdf
- See also: Centro Nacional de Epidemiología. CIBERESP. Instituto de Salud Carlos III. Informe epidemiológico sobre la situación del Herpes Zóster en España. [Internet]. 2020. [Consultado 18 Feb 2024]. — https://www.isciii.es/QueHacemos/Servicios/VigilanciaSaludPublicaRENAVE/EnfermedadesTransmisibles/Documents/archivos%20A-Z/HERPES%20ZOSTER/Informe_HZ_Espa%C3%B1a_1998-2018.pdf
- See also: Patkia A., Vorab A., Parikh R., Kolhapure S., Agrawal A., Dash R. Herpes zoster in outpatient departments of healthcare centers in India: a review of literatura. Human vaccines&immunotherapeutics. [Internet]. 2021. [Consultado 29 Mar 2024]. — https://pubmed.ncbi.nlm.nih.gov/34520327/
- See also: Ralph Tayyar R., Ho D. Herpes Simplex Virus and Varicella Zoster Virus Infections in Cancer Patients. Viruses. [Internet]. 2023. [Consultado 28 Mar 2024];15, 439. — https://pubmed.ncbi.nlm.nih.gov/36851652/
- See also: Van Oorschot D., McGirr A., Goulet P., Koochaki P., Pratiwadi R., Shah S., Curran D. A Cross-Sectional Concept Elicitation Study to Understand the Impact of Herpes Zoster on Patients' Health-Related Quality of Life. InfectDisTher. [Internet]. 2022. — https://pubmed.ncbi.nlm.nih.gov/34994924/
- See also: Sollie M., Jepsen P., Sørensen, JA. (2022). Patient-reported quality of life in patients suffering from acute herpes zoster-a systematic review with meta-analysis. British journal of pain. [Internet]. 2022. [Consultado 28 Mar 2024]; 15 16(4), 404-419. — https://pubmed.ncbi.nlm.nih.gov/36032345/
- See also: Díez Domingo J., Curran D., Cambronero MR., Garcia Martinez JA., Matthews S. Economic Burden and Impact on Quality of Life of Herpes Zoster in Spanish Adults Aged 50 Years or Older: A Prospective Cohort Study. Advances in therapy. [Internet]. 2021. [C — https://pubmed.ncbi.nlm.nih.gov/34013498/
- See also: Matthews S., De Maria A., Passamonti M.,Ristori G., Loiacono I., Puggina A., Curran D. The Economic Burden and Impact on Quality of Life of Herpes Zoster and Postherpetic Neuralgia in Individuals Aged 50 Years or Older in Italy. Open ForumInfectDis. [ — https://pubmed.ncbi.nlm.nih.gov/30793003/
- See also: Zhao D, Suo L., Lu L., Pan J., Peng X., Wang Y., Pang X. Impact of herpes zoster and post-herpetic neuralgia on health-relate. Vaccine X. [Internet]. 2023. [Consultado 28 Mar 2024]; 15, 100415. — https://pubmed.ncbi.nlm.nih.gov/38124774/
- See also: Curran D., Hunjan M., El Ghachi A., El-Hahi Y., Bianco V., Ferreira G. Herpes zoster related healthcare burden and costs in immunocompromised (IC) and IC-free populations in England: an observational retrospective database analysis. BMJ Open. [Interne — https://pubmed.ncbi.nlm.nih.gov/31462457/
- See also: Chen L., Li J., Liu H., Yang P., Zuo Y., Ye L. Interventions for zoster-associated pain: A retrospective study based on the clinical database.Front Neurol. [Internet]. 2022. [Consultado 29 Mar 2024];13:1056171. — https://pubmed.ncbi.nlm.nih.gov/36504661/
- See also: Lin CS., Lin YC., Lao HC., Chen CC. Interventional Treatments for Postherpetic Neuralgia: A Systematic Review. Pain Physician. [Internet]. 2019. [Consultado 28 Mar 2024]; 22,209-228. — https://pubmed.ncbi.nlm.nih.gov/31151330/
- See also: Zeng F., Wang M., Zhang D. Cost-effectiveness analysis of 5% lidocaine-medicated plaster compared with pregabalin for the treatment of post-herpetic neuralgia in China.Pain and therapy. [Internet]. 2021. [Consultado 30 Mar 2024]; 10(1), 675-689. — https://pubmed.ncbi.nlm.nih.gov/33894728/
- See also: Sollie M., Jepsen P., Sorensen JA. Patient-reported quality of life in patients suffering from acute herpes zoster-a systematic review with meta-analysis. British Journal of Pain. [Internet]. 2022. [Consultado 18 Feb 2024]; 16(4) 404-419. — https://pubmed.ncbi.nlm.nih.gov/36032345/
- See also: Hideo Hashizumea H., NakataniaE. ,Satoa Y., Gotoc H. , Yagic H., Miyachi Y. A new susceptibility index to predict the risk of severe herpes zoster-associated pain: A Japanese regional population-based cohort study, the Shizuoka study. Journal of Derma — https://pubmed.ncbi.nlm.nih.gov/35181196/
- See also: Centro Nacional de Epidemiología. CIBERESP. Instituto de Salud Carlos III. Informe epidemiológico sobre la situación del Herpes Zóster en España. [Internet]. Madrid; 2020. [Consultado 18 Feb 2024]. — https://www.isciii.es/QueHacemos/Servicios/VigilanciaSaludPublicaRENAVE/EnfermedadesTransmisibles/Documents/archivos%20A-Z/HERPES%20ZOSTER/Informe_HZ_Espa%C3%B1a_1998-2018.pdf
- See also: Sicras-Mainar A., Navarro-Artieda R., Ibanez-Nolla J., Perez-Ronco J. Incidence, resource use and costs associated with postherpetic neuralgia: a population-based retrospective study. Rev Neurol. . [Internet].2012[Consultado 10 Abr 2024]; 55:449-461. — https://pubmed.ncbi.nlm.nih.gov/23055426/